CLINICAL TRIAL: NCT01492270
Title: PICTURE - Prostate Imaging (Multi-parametric MRI and Prostate HistoScanning™) Compared to Transperineal Ultrasound Guided Biopsy for Significant Prostate Cancer Risk Evaluation.
Brief Title: Imaging for Significant Prostate Cancer Risk Evaluation
Acronym: PICTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: Advanced Medical Diagnostics s.a. (Industry)
Responsible Party: Principal Investigator, Professor Mark Emberton, Professor of Interventional Oncology, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11/LO/1657
Record Dates: First submitted 2011-12-06; First posted 2011-12-14 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Multi parametric MRI; Prostate HistoScanning; Transperineal prostate mapping biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Image-Guided Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prostate HistoScanning — Advanced Ultrasound assessment of the prostate
Procedure: Multi-parametric MRI — Multi-sequence Magnetic resonance imaging of the prostate
Procedure: Transperineal prostate mapping biopsy — Needle biopsy of the perineum via the transperineal route at 5mm intervals guided by the use of ultrasound.
Procedure: Image guided biopsies — Biopsies targeted to lesions seen at a) Prostate HistoScanning and b) mp-MRI. In men with an MRI lesion further MRI/US registration biopsies will be obtained
  Other Names: Targeted Biopsy

SUMMARY:
The incidence of prostate cancer is rising however the number of deaths from prostate cancer is stable. Meaning the investigators are diagnosing many men with prostate cancer that will not impact on their life. The rise in incidence is mainly due to increased use of the blood test Prostate Specific Antigen (PSA), as a screening test.

Currently men suspected of having prostate cancer, identified by a raised PSA undergo trans-rectal ultrasound guided prostate biopsy (TRUS biopsy). Many men have this test unnecessarily, only 1/3 being diagnosed with prostate cancer. TRUS biopsy is problematic as it is random and performed blind-the operator does not know where the cancer is. Thus many low-risk cancers that do not need treating are diagnosed and many high risk cancers are missed or incorrectly classified. So, men with a negative biopsy or those with low risk disease are usually advised to undergo another TRUS biopsy.

An imaging test is needed that could help men and their doctors decide whether the biopsy is a true reflection of what is inside his prostate.

The investigators will test the role of two imaging tests. The first, multi-parametric magnetic resonance imaging (mp-MRI) uses magnetic signals from the body to form images. The second, Prostate HistoScanning™ (PHS) uses sound-waves. The investigators will compare the results of these tests with a detailed biopsy map-transperineal template prostate mapping biopsy (which is currently the best way to find out what is in the prostate but requires multiple biopsies to be taken under general anaesthetic. Eligible men will have undergone one or more TRUS biopsies and who have been advised to have further tests on as part of standard of care. They will be recruited from UCLH referral letters and clinics.

The investigators aim is to see if either of these tests can confidently rule out the presence of clinically important disease.

ELIGIBILITY:
Inclusion Criteria:

* Men who have undergone prior trans-rectal biopsies.
* Men undergoing further evaluation of their prostate and who are seeking characterisation using Transperineal Template Prostate Mapping Biopsy.

Exclusion Criteria:

* Previous history of prostate cancer treatment
* Men unable to have MRI scan, or in whom artefact would reduce quality of MRI.
* Men unable to have general or regional anaesthesia
* Men unable to give informed consent

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of men who could avoid repeat biopsy as determined by the Negative predictive value and specificity of mp-MRI for Clinically significant disease. | 18 months
  Performance characteristics of mp-MRI for ruling out CLINICALLY SIGNIFICANT prostate cancer as determined by negative predictive value and specificity
Number of men who could avoid repeat biopsy as determined by the negative predictive value and specificity of Prostate HistoScanning for Clinically significant disease. | 18 months
  Performance characteristics of Prostate HistoScanning for ruling out CLINICALLY SIGNIFICANT prostate cancer as determined by negative predictive value and specificity

SECONDARY OUTCOMES:
Proportion of men correctly identified as having no cancer on Imaging (mp-MRI and Prostate HistoScanning) | 18 months
  Negative predictive value of Imaging compared to Transperineal template Mapping prostate biopsy.
Number of men correctly identified by Imaging (mp-MRI and Prostate HistoScanning) to have CLINICALLY SIGNIFICANT disease | 18 months
  Number of men correctly identified by each test to have clinically significant disease as detected by Transperineal Template Mapping Biopsy
Test- retest reproducibility of Prostate HistoScanning™. | 18 months
  The reproducibility of Prostate HistoScanning will be assessed by looking at the predicted cancer volume and location of the HistoScanning investigation at two time points.
Proportion of patients with correct disease risk stratification using MRI/US guided biopsies as determined by sensitivity and specificity | 18 months
  Performance characteristics of MRI/US registration targeted biopsies compared to i) systematic biopsies and ii) cognitive targeted biopsies in prostate cancer risk stratification as determined by sensitivity and specificity
Number of patients with bothersome Lower Urinary tract symptoms following Transperineal Template Mapping biopsy | 18 months
  Assessment of alterations in Lower Urinary tract function following Transperineal Template Mapping Biopsy
  IPSS, IPSS-QoL, Continence Function Questionnaire.
Number of patients with worsened erectile function compared to baseline following Transperineal Template Mapping biopsy | 18 months
  Assesment of erectile function compared to baseline will be made using questionnairres.
  IIEF

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MBBS,MD,FRCS, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospitals, London, London, United Kingdom

REFERENCES:
- [Derived] Simmons LAM, Kanthabalan A, Arya M, Briggs T, Charman SC, Freeman A, Gelister J, Jameson C, McCartan N, Moore CM, van der Muelen J, Emberton M, Ahmed HU. Prostate Imaging Compared to Transperineal Ultrasound-guided biopsy for significant prostate cancer Risk Evaluation (PICTURE): a prospective cohort validating study assessing Prostate HistoScanning. Prostate Cancer Prostatic Dis. 2019 May;22(2):261-267. doi: 10.1038/s41391-018-0094-1. Epub 2018 Oct 2. PMID 30279583
- [Derived] Simmons LAM, Kanthabalan A, Arya M, Briggs T, Barratt D, Charman SC, Freeman A, Hawkes D, Hu Y, Jameson C, McCartan N, Moore CM, Punwani S, van der Muelen J, Emberton M, Ahmed HU. Accuracy of Transperineal Targeted Prostate Biopsies, Visual Estimation and Image Fusion in Men Needing Repeat Biopsy in the PICTURE Trial. J Urol. 2018 Dec;200(6):1227-1234. doi: 10.1016/j.juro.2018.07.001. Epub 2018 Jul 11. PMID 30017964
- [Derived] Miah S, Eldred-Evans D, Simmons LAM, Shah TT, Kanthabalan A, Arya M, Winkler M, McCartan N, Freeman A, Punwani S, Moore CM, Emberton M, Ahmed HU. Patient Reported Outcome Measures for Transperineal Template Prostate Mapping Biopsies in the PICTURE Study. J Urol. 2018 Dec;200(6):1235-1240. doi: 10.1016/j.juro.2018.06.033. Epub 2018 Jun 27. PMID 29940251